CLINICAL TRIAL: NCT05478265
Title: Patient Observational Pain and Activity Survey (POPAS) Study Using RS-4i Sequential Stimulator With Intersperse Technology in Axial Spine and Peripheral Joint Pain
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, David Majors, Principal Investigator, University of California, Irvine
Other Study IDs: 20216774
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (6):
- Axial Spine only, Age 65+
  Interventions: Device: RS-4i Plus
- Axial Spine only, Age 18-64
  Interventions: Device: RS-4i Plus
- Peripheral Joint only, Age 65+
  Interventions: Device: RS-4i Plus
- Peripheral Joint only, Age 18-64
  Interventions: Device: RS-4i Plus
- Axial + Peripheral Joint, Age 65+
  Interventions: Device: RS-4i Plus
- Axial + Peripheral Joint, Age 18-64
  Interventions: Device: RS-4i Plus

INTERVENTIONS:
Device: RS-4i Plus — RS-4i Plus in an FDA-regulated prescription TENS medical device that outputs and INF signal and a NMES signal and Intersperse signal, which combines INF and NMES into a single treatment.

SUMMARY:
Spine pain and joint pain are among the most common worldwide ailments and directly contributes to disability as well as increased duration of care. Spine and joint pain affect work sick leave, production and increased financial costs to healthcare. Non-invasive treatments for spine and joint pain can vary widely from lifestyle changes, physical therapy, oral medication, and select medical devices, that can improve pain level and help improve the quality of life of individuals. Thus, the general population suffers from an ailment that has multiple conservative treatment options with variable outcomes.

Transcutaneous Electrical Neuromuscular Stimulation (TENS) has been show to decrease pain and restore function. Interferential therapy (INF) is a specific signal type that is effective for reducing musculoskeletal pain. Neuromuscular Electrical Stimulation (NMES) uses a specific signal type to cause muscles to contract and therefore provide functional improvement. The RS-4i Plus is an FDA-regulated prescription TENS medical device that outputs an INF signal and a NMES signal, and a unique Intersperse signal, which combines NMES and INF into a single treatment. Therefore, the goal of this study is to determine if use of the prescribed RS-4i Plus in patients presenting with pain, axial or peripheral joint, can be efficacious in decreasing the patient's pain and improving their activity measured at one month, three months, and six months of use.

ELIGIBILITY:
Inclusion Criteria:

1. chronic and persistent MSK lumbar back pain for greater than 12 weeks as documented in patient records
2. Age 18 to 89
3. Willingness to comply with study protocol
4. Signed Patient Consent on file
5. Verified patient usage collected from RS-4i Plus via patient data adapter

Exclusion Criteria:

1. Pregnancy
2. Any contraindications, as indicated in the RS-4i Plus prescribing information
3. Substantial allergy to adhesives
4. Skin infection or irritation of skin where electrodes are to be placed
5. Pacemaker/ICD
6. Abnormal skin sensation
7. Serious psychological disorder
8. End-stage cardiac, peripheral arterial or pulmonary disease
9. h/o recent vertebral fracture
10. Severe degenerative or traumatic neuromuscular disease
11. Non-English speaking
12. Uncontrolled diabetes meelitus (Hb A1c> 8.5%)
13. ESRD or ESHD
14. Active cancer

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be current adult patients of the UCI PM&R or Orthopedic Department
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Level of Pain / Function using NRS | 1 month
  Outcome with be rated on a scale of 0-10, in which 10 is the most severe pain / worst function and 0 is the least pain / best function. The time frame will include assessment at 1 month interval to determine if the intervention is showing a change / long term improvement in the pain / function
Level of Pain / Function using NRS | 3 month
  Outcome with be rated on a scale of 0-10, in which 10 is the most severe pain / worst function and 0 is the least pain / best function. The time frame will include assessment at 3 month interval to determine if the intervention is showing a change / long term improvement in the pain / function
Level of Pain / Function using NRS | 6 months
  Outcome with be rated on a scale of 0-10, in which 10 is the most severe pain / worst function and 0 is the least pain / best function. The time frame will include assessment at 6 month interval to determine if the intervention is showing a change or long term improvement in the pain / function

CONTACTS AND LOCATIONS:
Locations (1):
- University of California at Irvine Medical Center, Orange, California, United States